CLINICAL TRIAL: NCT04206800
Title: Effect of Ejaculatory Abstinence on Semen Parameters in Male Factor Infertility Patients: a Randomized Controlled Study
Brief Title: Effect of Ejaculatory Abstinence on Semen Parameters in Male Factor Infertility Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling participants
Sponsor: Boston IVF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P001037
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Infertility, Male
Keywords: in-vitro fertilization; total motile sperm; male infertility; ejaculatory abstinence
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (No Intervention): Routine care is normally having men abstain from ejaculation from 2 to 5 days prior to the scheduled oocyte retrieval date. Men in the routine care arm will abstain from ejaculation greater than 48 hours before providing a semen sample the day of the scheduled oocyte retrieval.
- Ejaculatory abstinence less than 24 hours (Experimental): Males will ejaculate within 24 hours of the scheduled oocyte retrieval date.
  Interventions: Diagnostic Test: Ejaculatory abstinence less than 24 hours

INTERVENTIONS:
Diagnostic Test: Ejaculatory abstinence less than 24 hours — Males will have ejaculatory abstinence less than 24 hours before providing a semen sample the day of egg retrieval
  Arms: Ejaculatory abstinence less than 24 hours

SUMMARY:
The purpose of this study is to compare semen parameters with in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) when male factor infertility patients abstain from ejaculation more than 48 hours (routine care) or less than 24 hours from the day of the partner's oocyte retrieval. The investigators hypothesize that total motile sperm count will be improved with ejaculatory abstinence (EA) less than 24 hours. Information from this trial could allow investigators to optimize chances for a successful pregnancy in patients who need IVF/ICSI.

DETAILED DESCRIPTION:
Overview This will be a randomized controlled study to compare semen parameters following EA for more than 48 hours (routine care) or less than 24 hours from the day of the partner's oocyte retrieval among male factor infertility patients who receive IVF/ICSI.

Methods Study participation will not influence any element of IVF treatment and all participants will be receiving the standard of care at Boston IVF. For participants who meet eligibility criteria and provide informed verbal consent, baseline demographic data will be obtained from the medical record including for example: age, race, education level, height, weight, baseline semen analysis, testosterone level, follicle stimulating hormone (FSH) level. Demographic data on the female partner will include parameters such as: age, race, education level, height, weight, gravidity, parity, anti-mullerian hormone level, and day 3 FSH.

Eligible participants will have the study introduced by the medical care team. Eligible participants will be given information on study details as well as an ejaculatory calendar/survey that can be used if the participant enrolls in the study. The medical care team will inform eligible participants that participants will receive a recruitment email from the research team at BIVFresearch@bostonivf.com followed by a phone call from the research team to see if eligible participants are willing to participate. Eligible participants who meet inclusion and exclusion criteria whom do not get information regarding the study from the medical care team will also receive a recruitment email. A research member will call eligible participants to obtain verbal consent to enroll in the study. If the participant does not answer, a voicemail will be recorded followed by a second phone call the following day. The recruitment email and verbal consent will occur between the pre-IVF period and before stimulation day 4 of the IVF cycle. If a participant consents to enrollment, the investigators will make a note in the treatment plan for the partner's IVF cycle. Enrolled participants will receive a phone call from a member of the research team during stimulation day 6 to 8 to randomize the participant to EA greater than 48 hours (routine care) or EA less than 24 hours from the day of the partner's oocyte retrieval. If the participant does not answer, a voicemail will be recorded followed by a second phone call the following day.

The semen sample provided on day of oocyte retrieval will be analyzed with a basic and advanced semen panel. Any remaining samples will be discarded per routine practice. Prior to providing the semen sample, participants will turn in the completed survey/ejaculation history calendar to a member of the research team. Blank copies will be available for participants the day of oocyte retrieval if needed.

There is no clinical risk to the IVF cycle as the procedures followed are standard clinical practice. Study participation will not influence any element of the IVF treatment except for EA counseling. Currently, there is no set protocol on how EA counseling is performed. Counseling on EA varies among the medical care teams at Boston IVF as some patients may or may not receive explicit EA instructions. Patients may be counseled by the medical care team with recommendations to abstain for greater than 48 hours. All participants in the study will use ICSI to fertilize eggs and the number of sperm needed for treatment will not be compromised by ejaculatory abstinence less than 24 hours. Participants who crossover to the alternate treatment arm will continue participation in the study so that investigators can collect cycle outcome data. IVF stimulation protocols will be according to standard practice. ICSI and embryology practice will follow standard practice. Selection of embryos will be based on the current embryology laboratory selection protocols or by preimplantation genetic testing for aneuploidy (PGT-A). The number of embryos transferred will be based on the usual American Society of Reproductive Medicine guidelines. Any unused embryos will be disposed of or cryopreserved per standard clinical protocols.

Intervention Participants will be randomized to EA more than 48 hours (routine care) or less than 24 hours from the day of the partner's oocyte retrieval.

Randomization The investigators will use computer-generated block randomization in REDCap to randomize participants in a 1:1 ratio to the EA period more than 48 hours (routine care) or less than 24 hour. Randomization will be stratified by whether the participants receive PGT-A. The investigators will call participants on stimulation day 6 to 8 to notify which treatment arm the participant was randomized to. The participant can withdraw from the study at any time if desired or will have an opportunity to not continue with the treatment arm the participant was randomized to. The investigators anticipate that most of the crossovers will occur due to participants wishing to be in the alternate EA period or not being able to produce a sample in the window assigned.

Sample Size Justification The sample size calculation is based on data from Boston IVF from 2013 to 2018 for patients with less than 3 million total motile sperm post prep for IVF/ICSI patients. The mean percentage of total motile sperm is 38% ± 24 which will be the investigators control group. The investigators hypothesize that the mean percentage of total motile sperm at the time of oocyte retrieval will increase to 48. In order to achieve 80% power to detect the specified difference using a two-sided alpha of 0.05, the investigators will need 90 evaluable participants per arm. The investigators anticipate that approximately 15% of participants will drop out, and the investigators will inflate the sample size by another 15% to account for a non-normal distribution. Thus, the investigators aim to randomize 117 participants per arm for a total of 234 participants.

Data Analysis Descriptive data will be presented as a proportion, mean with standard deviation or median with interquartile range. Comparisons will be made using Chi-square or Fisher's exact test for categorical variables and parametric or non-parametric tests for continuous variables based on data distribution. Log-binomial regression will be used to estimate risk ratios and 95% confidence intervals for the primary and secondary outcomes. While the investigators anticipate that randomization will balance the distribution of measured and unmeasured potential confounders in the two study arms, if this is not the case, the investigators will assess the influence of potential confounders as needed. All data will be analyzed with SAS 9.4 (SAS Institute Inc., Cary, NC, USA). All tests will be two sided and a P value <0.05 will be required to confer significance.

ELIGIBILITY:
Inclusion Criteria:

* Male Age 18 - 50 years and female age < 38 years
* First IVF cycle
* Abnormal semen parameters (at least 1 of the following on 2 semen analysis with at least one being in the past 12 months): a) sperm concentration < 10 million/mL; b) unprocessed semen analysis with < 10 million motile sperm or processed semen analysis with < 3 million motile sperm; c) < 2 % normal forms (strict Kruger morphology)
* Female AMH > 0.7 and/or and day 2-4 FSH < 12

Exclusion Criteria

* Donor sperm
* Males with less than 200,000/mL sperm in the ejaculate
* Utilization of a gestational carrier
* Frozen donor egg
* Female morbid obesity: BMI > 40
* History of recurrent pregnancy loss (≥2 spontaneous abortions)
* Preimplantation genetic testing - (M or SR) Monogenetic disorders or chromosomal rearrangement
* The use of non-ejaculated sperm (testicular sperm extraction)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Penzias, MD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Care | Ejaculatory Abstinence Less Than 24 Hours
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care | Ejaculatory Abstinence Less Than 24 Hours | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (2.74) | 32 (0) | 35.2 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Motile Sperm (Million)
Description: total motile sperm (million sperm) is calculated from the semen analysis by calculating: volume x concentration x motility. This gives the total motile sperm value. The difference in total motile sperm was calculated from the participants baseline semen analysis (previous analysis before starting IVF treatment) to the semen analysis the day of the egg retrieval. The mean calculated can be interpreted as a decrease (change) in total motile sperm from the participants baseline semen analysis to the semen analysis the day of the egg retrieval.
Time Frame: Change in baseline and 1-5 months
Measure: Mean (Standard Deviation); unit: million sperm
Arm/Group | Routine Care | Ejaculatory Abstinence Less Than 24 Hours
Number analyzed (Participants) | 4 | 1
million sperm | 14.86 (24.99) | 7.94 (0)

2. Secondary Outcome: Live Birth Rate
Description: defined as delivery > 23 weeks gestation
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Fertilization Rate
Description: Number of fertilized eggs per oocyte retrieved
Time Frame: 18 hours after insemination
Reporting Status: Not Posted

4. Secondary Outcome: Embryo Development
Description: Asses the rate of embryo development
Time Frame: up to 7 days post egg retrieval
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Pregnancy Rate
Description: defined as confirmation of gestational sac on ultrasound
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Miscarriage Rate
Description: miscarriages per total number of pregnancies
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Ongoing Pregnancy Rate
Description: defined as confirmation of a gestational sac with at least one fetal pole with a fetal heartbeat
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Semen Analysis
Description: Changes in semen analysis from baseline diagnostic sample, an advanced semen analysis panel
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted

9. Secondary Outcome: Preimplantation Genetic Testing
Description: number of euploid and aneuploid embryos (if preimplantation genetic testing-aneuploidy [PGT-A] performed)
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Protocols were already standard of care
Arm/Group | Routine Care | Ejaculatory Abstinence Less Than 24 Hours
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04206800/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04206800/ICF_001.pdf